CLINICAL TRIAL: NCT04501003
Title: Investigation of Implantation Markers of Anomalies Classified as U1-A Uterine According to ESHRE/ESGE Classification of Female Genital Tractus Anomalies in Biopsy Specimens Obtained From the Lateral Walls of the Endometrium
Brief Title: Investigation of U1-A Uterine Anomalies Implantation Markers From the Lateral Walls of the Endometrium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Sezin Oral Yıldız, Resident, Ufuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1/190/2019
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: T-Shaped Uterus; Infertility, Female; Genital Tract Anomalies
Keywords: T-Shaped Uterus; Infertility, Female; Intregrin Beta 3; Genital Tract Anomalies
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bipolar cutting electrode (26040 BL1 Karl Storz, Tuttlingen) (Other): With the bipolar cutting electrode (26040 BL1 Karl Storz, Tuttlingen. Germany), a single incision was made from the bottom of the ostium onto the lateral walls up to the isthmus, with both lateral horns perpendicular to myometrium. The depth of the incision was between 5 and 7 mm.
  Interventions: Device: Bipolar cutting electrode (26040 BL1 Karl Storz, Tuttlingen)

INTERVENTIONS:
Device: Bipolar cutting electrode (26040 BL1 Karl Storz, Tuttlingen) — With the bipolar cutting electrode (26040 BL1 Karl Storz, Tuttlingen. Germany), a single incision was made from the bottom of the ostium onto the lateral walls up to the isthmus, with both lateral horns perpendicular to myometrium. The depth of the incision was between 5 and 7 mm. The cavity was widened to be triangular and symmetrical. Both tubal ostium surgeries were clearly observed at the end of the surgery. All patients were discharged on the day of surgery and no hormonal therapy and intrauterine balloon was applied after surgery. Approximately 3 months after the hysteroscopic T-shaped operation, an office hysteroscopy operation was planned to control patients in the secretory phase, to perform uterine cavity and post-operative fly control and to receive post-operative control endometrial biopsy specimens.

SUMMARY:
Various types and classes of uterine malformations have been identified and the ESHRE / ESGE classification system has recently been published on female genital system anomalies. Postoperative positive pregnancy results were obtained in studies conducted in patients with infertility, recurrent implantation failure, and recurrent pregnancy loss, which were not previously described in T-shaped uterine anomalies. Considering the increase in endometrial gland and vascularity after the surgical procedure performed in these patients, our primary goal in our study is to compare the number of implantation markers (αVβ3 integrin) and subepithelial glands in the specimen biopsies taken from the lateral walls of the endometrium before and after hysteroscopic surgery in patients with class U1a anomalies.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 age,
2. Have no systemic disease,
3. ESGE U1-A having uterine anomaly,
4. Primary infertile, recurrent implantation loss, recurrent pregnancy loss history,
5. Not having previous uterine surgery.

Exclusion Criteria:

1. Patients over the age of 45 under the age of 18,
2. Those with systemic disease (Hypertension, Heart Disease, Asthma, Renal Disease, Liver Disease, Epilepsy),
3. Having previous uterine surgery,
4. Those who gave birth.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of endometrial lateral wall biopsies before and after hysteroscopic metroplasty in patients with T-shaped uterus. | Baseline
  From the endometrium biopsies taken before and after the operation, the implantation marker beta 3 integrin was examined to determine if there was any change in the implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Chan YY, Jayaprakasan K, Zamora J, Thornton JG, Raine-Fenning N, Coomarasamy A. The prevalence of congenital uterine anomalies in unselected and high-risk populations: a systematic review. Hum Reprod Update. 2011 Nov-Dec;17(6):761-71. doi: 10.1093/humupd/dmr028. Epub 2011 Jun 24. PMID 21705770
- [Background] Grimbizis GF, Gordts S, Di Spiezio Sardo A, Brucker S, De Angelis C, Gergolet M, Li TC, Tanos V, Brolmann H, Gianaroli L, Campo R. The ESHRE/ESGE consensus on the classification of female genital tract congenital anomalies. Hum Reprod. 2013 Aug;28(8):2032-44. doi: 10.1093/humrep/det098. Epub 2013 Jun 14. PMID 23771171
- [Background] Valle RF, Ekpo GE. Hysteroscopic metroplasty for the septate uterus: review and meta-analysis. J Minim Invasive Gynecol. 2013 Jan-Feb;20(1):22-42. doi: 10.1016/j.jmig.2012.09.010. PMID 23312243
- [Background] Paradisi R, Barzanti R, Fabbri R. The techniques and outcomes of hysteroscopic metroplasty. Curr Opin Obstet Gynecol. 2014 Aug;26(4):295-301. doi: 10.1097/GCO.0000000000000077. PMID 24978851
- [Background] Giacomucci E, Bellavia E, Sandri F, Farina A, Scagliarini G. Term delivery rate after hysteroscopic metroplasty in patients with recurrent spontaneous abortion and T-shaped, arcuate and septate uterus. Gynecol Obstet Invest. 2011;71(3):183-8. doi: 10.1159/000317266. Epub 2010 Dec 11. PMID 21150155
- [Background] Fox NS, Roman AS, Stern EM, Gerber RS, Saltzman DH, Rebarber A. Type of congenital uterine anomaly and adverse pregnancy outcomes. J Matern Fetal Neonatal Med. 2014 Jun;27(9):949-53. doi: 10.3109/14767058.2013.847082. Epub 2013 Nov 26. PMID 24050215
- [Background] Bendifallah S, Faivre E, Legendre G, Deffieux X, Fernandez H. Metroplasty for AFS Class V and VI septate uterus in patients with infertility or miscarriage: reproductive outcomes study. J Minim Invasive Gynecol. 2013 Mar-Apr;20(2):178-84. doi: 10.1016/j.jmig.2012.11.002. Epub 2013 Jan 11. PMID 23317507
- [Background] Kaufman RH, Binder GL, Gray PM Jr, Adam E. Upper genital tract changes associated with exposure in utero to diethylstilbestrol. Am J Obstet Gynecol. 1977 May 1;128(1):51-9. doi: 10.1016/0002-9378(77)90294-0. PMID 851159
- [Background] Katz Z, Ben-Arie A, Lurie S, Manor M, Insler V. Beneficial effect of hysteroscopic metroplasty on the reproductive outcome in a 'T-shaped' uterus. Gynecol Obstet Invest. 1996;41(1):41-3. doi: 10.1159/000292033. PMID 8821883
- [Background] Garbin O, Ohl J, Bettahar-Lebugle K, Dellenbach P. Hysteroscopic metroplasty in diethylstilboestrol-exposed and hypoplastic uterus: a report on 24 cases. Hum Reprod. 1998 Oct;13(1O):2751-5. doi: 10.1093/humrep/13.10.2751. PMID 9804225
- [Background] Barranger E, Gervaise A, Doumerc S, Fernandez H. Reproductive performance after hysteroscopic metroplasty in the hypoplastic uterus: a study of 29 cases. BJOG. 2002 Dec;109(12):1331-4. doi: 10.1046/j.1471-0528.2002.01448.x. PMID 12504966
- [Background] de los Santos MJ, Mercader A, Galan A, Albert C, Romero JL, Pellicer A. Implantation rates after two, three, or five days of embryo culture. Placenta. 2003 Oct;24 Suppl B:S13-9. doi: 10.1016/s0143-4004(03)00172-3. PMID 14559025
- [Background] Tan BK, Vandekerckhove P, Kennedy R, Keay SD. Investigation and current management of recurrent IVF treatment failure in the UK. BJOG. 2005 Jun;112(6):773-80. doi: 10.1111/j.1471-0528.2005.00523.x. PMID 15924536
- [Background] Urman B, Yakin K, Balaban B. Recurrent implantation failure in assisted reproduction: how to counsel and manage. A. General considerations and treatment options that may benefit the couple. Reprod Biomed Online. 2005 Sep;11(3):371-81. doi: 10.1016/s1472-6483(10)60846-2. PMID 16176681
- [Background] Aflatoonian A, Baradaran Bagheri R, Hosseinisadat R. The effect of endometrial injury on pregnancy rate in frozen-thawed embryo transfer: A randomized control trial. Int J Reprod Biomed. 2016 Jul;14(7):453-158. PMID 27525329
- [Background] Dey SK, Lim H, Das SK, Reese J, Paria BC, Daikoku T, Wang H. Molecular cues to implantation. Endocr Rev. 2004 Jun;25(3):341-73. doi: 10.1210/er.2003-0020. PMID 15180948
- [Background] Lessey BA. Two pathways of progesterone action in the human endometrium: implications for implantation and contraception. Steroids. 2003 Nov;68(10-13):809-15. doi: 10.1016/j.steroids.2003.09.004. PMID 14667972
- [Background] Achache H, Revel A. Endometrial receptivity markers, the journey to successful embryo implantation. Hum Reprod Update. 2006 Nov-Dec;12(6):731-46. doi: 10.1093/humupd/dml004. Epub 2006 Sep 18. PMID 16982667